CLINICAL TRIAL: NCT06837610
Title: Inverted T Trabeculectomy for Primary Congenital Glaucoma, A Novel Technique
Brief Title: Inverted T Trabeculectomy Primary Congenital Glaucoma
Acronym: Inverte T trab
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelzaher Awwad, Dr, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inverted T trab PCG
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Glaucoma, Congenital, Surgical Treatment
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Retrospective, non-controlled case series
Masking Description: purposefully concealing treatment assignment to prevent outcomes from being influenced by biases due to knowledge of that assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary congenital glaucoma surgey (Other): Compare the Novel inverted T technique to the classic trabeculectomy in treatment of primary congenital glaucoma
  Interventions: Procedure: Inverted T trabeculectomy

INTERVENTIONS:
Procedure: Inverted T trabeculectomy — * Fornix-based conjunctival incision along with the opening of Tenon's capsule and dissection along the area of the potential bleb.
  * A 4 x 4 mm limbal-based scleral flap was fashioned using a crescent knife. Dissection was carried out up to the clear cornea.
  * A longitudinal tunnel was made through the scleral bed, starting from the limbus and extending 1 mm beyond the end of the scleral flap. Afterwards, the horizontal limb of the Inverted T was created. (Figure 2)
  * A paracentesis was made using an MVR blade.
  * The anterior chamber was entered using an MVR blade. Kelly's punch was used to excise 1.5 x 1.5 mm of scleral bed at the limbus at the base of the vertical limb of the figure (T), and then a peripheral iridectomy was performed using Vannas scissors.
  * The scleral flap was then closed using two fixed 10/0 Nylon sutures, one at each corner.

SUMMARY:
This study aims to evaluate the safety and efficacy of novel Inverted T trabeculectomy in Primary Congenital Glaucoma (PCG). It enrolled 50 eyes of 25 children with PCG. The mean age at the time of surgery was 12±11 months, and the mean presenting IOP was 40±4 mmHg. Patients with previous intra-ocular or conjunctival surgery, those who had significant ocular trauma, and patients with congenital glaucoma associated with ocular anomalies diseases were excluded from the study. All patients had Inverted T trabeculectomy under general anesthesia. The IOP in the operated eyes was followed up for 36 months.

DETAILED DESCRIPTION:
This study included patients from the glaucoma clinic at Benha University Hospital between April 2015 and October 2017. All were diagnosed with PCG based on an intraocular pressure (IOP) measurement of 21 mmHg or more at birth or shortly after, up to the age of 12 months. Patients with previous intraocular or conjunctival surgery, those with significant ocular trauma, and those with congenital glaucoma associated with other ocular anomalies that would affect IOP were excluded from the study.

The procedure principles and potential complications were discussed with the children's parents or legal guardians, and they gave written informed consent before surgery. This study was approved by the Benha Faculty of Medicine's ethical committee (Approval number RC 9-1-2025) and conducted according to Helsinki's declaration.

All patients underwent complete ophthalmic examination under general anaesthesia before surgery. IOP was measured 5 minutes after injecting intravenous Ketamine 1mg/kg for induction of anaesthesia. We used a Perkins tonometer (Haag-Streit, UK) to measure the IOP before applying the eyelid speculum. Corneal clarity was assessed under a surgical microscope, the corneal diameter was recorded using a surgical caliber, and fundus examination was done by indirect ophthalmoscope. A surgical Swan Jacob gonioprism assessed the anterior chamber angle when the cornea was clear enough to achieve a good view.

All surgeries were performed under general anaesthesia by the same surgeon (AEH).

ELIGIBILITY:
Inclusion Criteria:

* PCG based on an intraocular pressure (IOP) measurement of 21 mmHg or more at birth or shortly after, up to the age of 12 months

Exclusion Criteria:

* Patients with previous intraocular or conjunctival surgery, those with significant ocular trauma, and those with congenital glaucoma associated with other ocular anomalies that would affect IOP were excluded from the study

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Post op IOP | 18 months
  IOP lower than 21 mmHg or > 20% reduction from the baseline IOP in at least two consecutive follow-up visits without IOP-lowering medications and without vision-threatening complications

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Qualubia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The data supporting this study's findings are available from the corresponding author, upon reasonable request.